CLINICAL TRIAL: NCT03505801
Title: Confirm Rx Insertable Cardiac Monitor SMART Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10176
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrhythmias; Symptoms and Signs; Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Signs and Symptoms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Confirm Rx ICM insertion procedure — Insertion of Confirm Rx ICM device

SUMMARY:
The purpose of the Confirm Rx SMART Registry is to collect real world data to assess the safety and performance of the Confirm Rx Insertable Cardiac Monitor (ICM) and system over a 12 month period. A sub-set of subjects enrolled in the Confirm Rx SMART Registry will meet the Post Market Clinical Follow-Up (PMCF) requirement for CE mark.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication for continuous arrhythmia monitoring with an ICM
* Have a cellular phone or the ability or willing to use a St. Jude Medical mobile transmitter that is compatible with the MyMerlin App and able to communicate with the Confirm Rx ICM device.
* Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
* Are 18 years of age or older, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Subject is implanted with or indicated for implant with a pacemaker, implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy (CRT) device.
* Enrolled or intend to participate in a clinical drug and/or device study, which could confound the results of this trial as determined by the sponsor, during the course of this clinical study.
* Have a life expectancy of less than 1 year due to any condition.
* Have a previous ICM placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over the age of 18 years (or of legal age specific to state and national law) who experience unexplained symptoms such as: dizziness, palpitations, chest pain, syncope, and shortness of breath, as well as subjects who are at risk for cardiac arrhythmias, have been previously diagnosed with atrial fibrillation, or who are susceptible to developing atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 1826 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from device SADEs and serious procedure related SAEs | 1 month post insertion procedure

SECONDARY OUTCOMES:
Freedom from device SADEs and serious procedure related SAEs | 12 months post insertion procedure
R wave amplitude | 12 months post insertion procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Quartieri, MD, Principal Investigator — Arcispedale S. Maria Nuova - IRCCS l
Locations (113):
- United States (15):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Heart Clinics, Coeur d'Alene, Idaho
  - Iowa Heart Center, West Des Moines, Iowa
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Adventist HealthCare White Oak Medical Center, Silver Spring, Maryland
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
- Hôpital Central de l'Armée, Algiers, Algeria
- Argentina (2):
  - Instituto Argentino de Diagnostico y Tratamiento, Buenos Aires
  - Clinica Provincial, Merlo
- Austria (3):
  - Kepler Universitätsklinikum GmbH, Linz
  - Krankenhaus der Stadt St. Pölten, Sankt Pölten
  - Universitätsklinikum Tulln, Tulln
- Belgium (3):
  - Hopital Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - CHU Liège Sart Tilman, Liège
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Institut de Cardiologie de Quebec (Hospital Laval), Québec, Quebec
  - CHUM, Montreal
  - HSC, Eastern Health, St. John's
- Germany (16):
  - Asklepios Klinik St. Georg, Hamberg, Hamberg
  - Klinikum Idar-Oberstein GmbH, Idar-Oberstein, Hesse
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Klinikum Coburg GmbH, Coburg
  - Evangelisches Krankenhaus Kalk gGmbH, Cologne
  - Krankenhaus Porz am Rhein, Cologne
  - Medizinische Einrichtungen der Universität zu Köln, Cologne
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Klinikum Furth, Fürth
  - Klinikum Herford, Herford
  - Universitätsklinikum Leipzig AÖR, Leipzig
  - St.-Marien-Hospital GmbH, Lünen
  - München Grosshadern, München
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
- Semmelweis University, Budapest, Budapst, Hungary
- India (2):
  - Advance Medicare Research Institute (AMRI) Hospital, Dhakuria
  - Max Super Specialty Hospital, New Delhi
- Bnai Zion Medical Israel, Haifa, Haifa District, Israel
- Italy (9):
  - Azienda Ospedaliero Universitaria - Ospedali Riuniti Foggia, Foggia, Apulia
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - C.D.C. Citta di Aprilia, Aprilia
  - Az.Osp.Universitaria Consorziale Policlinico, Bari
  - Presidio Ospedaliero Giovan Battista Grassi, Ostia Antica
  - Casa di Cura Dpott. Pederzoli, Peschiera del Garda
  - Ospedale S. Andrea, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli di Roma, Roma
  - Policlinico Casilino, Roma
- Japan (9):
  - Yokohamashintoshi Neurosurgical Hospital, Yokohama, Kanagwa
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuok
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Akashi Medical Center, Hyōgo
  - St. Marianna University School of Medicine - Toyoko Hospital, Kawasaki
  - Kokura Memorial Hospital, Kitakyushu
  - University Hospital of Occupational & Environmental Health, Kitakyushu
  - Iwate Prefectural Central Hospital, Morioka
  - Osaka University Hospital, Suita
- Sabah Al-Ahmad Cardiac Centre, Kuwait City, Kuwait
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Netherlands (5):
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Martini Ziekenhuis, Groningen
  - Erasmus MC - Thoraxcenter, Rotterdam
  - Haga Ziekenhuis Locatie Leyenburg, The Hague
  - Maxima Medisch Centrum, Veldhoven
- Portugal (5):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar do Alto Ave, Unidade de Guimarães, Creixomil
  - Hospital de Santo Andre - Centro Hospitalar de Leiria, Leiria
  - Santa Maria Hospital, Lisbon
- Caribbean Heart Institute, Caguas, Puerto Rico
- Saudi Arabia (3):
  - King Fahad Armed Forces Hospital, Jeddah
  - King Abdullah Medical City in Holy Capital, Mecca
  - King Fahad Medical City, Riyadh
- Changi General Hospital, Singapore, Singapore, Singapore
- Slovakia (2):
  - Stredoslovenský ústav srdcových a cievnych chorôb, a.s., Banská Bystrica, Stredne
  - The National Institute of Cardiovascular Diseases, Bratislava
- South Africa (6):
  - Sunninghill Hospital, Johannesburg, Sandton
  - MedClinic Panorama, Cape Town, W Cape
  - Groote Schuur Hospital, Cape Town, W Cape
  - Unitas Hospital, Centurion
  - Busamed Hillcrest Private Hospital, Hillcrest
  - Busamed Gateway Private Hospital, Umhlanga
- South Korea (13):
  - Hallym University Sacred Heart Hospital, Anyang, Gyeongi
  - Inha University Hospital, Junggu, Gyeongi
  - Dong-A University Hospital, Busan, South Gyeongsang Province
  - Seoul National University Bundang Hospital, Seongnam, Sudogwn
  - Chung Ang University Hospital, Seoul, Sudogwn
  - Kosin University Gospel Hospital, Busan, Yeongnm
  - Ulsan University Hospital, Ulsan, Yeongnm
  - Keimyung University Dongsan Medical Center, Daegu
  - Asan Medical Centre, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Universitario de Badajoz, Badajoz, Extmdra
  - Hospital de Sant Joan Despí Moisès Broggi, Barcelona
  - Hospital Puerta de Hierro - Hospital Universitario, Majadahonda
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Alvaro Cunqueiro, Dept of EP & Arrhythmias, Vigo
- United Kingdom (3):
  - St. Thomas Hospital, London, London
  - Royal Bournemouth Hospital, Bournemouth
  - St Georges Hospital London, London

REFERENCES:
- [Derived] Quartieri F, Baek YS, Park JS, Kim TH, Honma K, Morimoto M, Kang KW, Feng L, Lee K, Grammatico A, Kaiser L. Continuing evaluation of atrial fibrillation detection after cryptogenic stroke: 2-year findings from a multicentre study with Confirm Rx ICM. Open Heart. 2025 Jun 12;12(1):e003242. doi: 10.1136/openhrt-2025-003242. PMID 40514061